CLINICAL TRIAL: NCT00000659
Title: A Phase II Trial of rsCD4 and AZT in Patients With AIDS or Advanced AIDS Related Complex (ARC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Biogen (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 133; C89-013-P
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 1990-07

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; Antigens, CD4; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — CD4 Antigens; Zidovudine

INTERVENTIONS:
Drug: CD4 Antigens
Drug: Zidovudine

SUMMARY:
Part 1A: To find the dose of zidovudine (AZT) that causes less than a 50 percent drop in HIV-1 p24 antigen levels in patients with AIDS and advanced AIDS related complex (ARC); to determine the pharmacokinetics (blood levels) of rsCD4 administered in combination with AZT. Parts 1B and 2: To test for additive or synergistic activity between rsCD4 and AZT as judged by falls in HIV-1 p24 antigen levels; and to evaluate the safety of rsCD4 and AZT in patients with AIDS and advanced ARC.

AZT has been shown to be effective in the treatment of AIDS and advanced ARC but not without toxicity. The most clinically significant toxicity is dose related inhibition of bone marrow function. Furthermore, HIV-1 isolates from patients treated for more than 6 months with AZT have now been found which appear to have reduced sensitivity to AZT. The incidence of toxicity and occurrence of virus with reduced sensitivity to AZT may result in the inability to administer AZT long-term to patients with AIDS and advanced ARC. Recombinant soluble CD4 (rCD4) has shown antiretroviral effects and has been shown to be safe when given to AIDS and ARC patients either as a single agent or in combination with AZT.

DETAILED DESCRIPTION:
AZT has been shown to be effective in the treatment of AIDS and advanced ARC but not without toxicity. The most clinically significant toxicity is dose related inhibition of bone marrow function. Furthermore, HIV-1 isolates from patients treated for more than 6 months with AZT have now been found which appear to have reduced sensitivity to AZT. The incidence of toxicity and occurrence of virus with reduced sensitivity to AZT may result in the inability to administer AZT long-term to patients with AIDS and advanced ARC. Recombinant soluble CD4 (rCD4) has shown antiretroviral effects and has been shown to be safe when given to AIDS and ARC patients either as a single agent or in combination with AZT.

Part 1A: Twenty p24+ patients with AIDS or advanced ARC are randomized to 4 dosing groups of 5 patients each. Patients are treated with AZT for 6 weeks at ranging doses to determine a minimally effective dose (MED). At the end of week 6, each patient is sequentially assigned to 1 of 5 groups of rCD4 / AZT combination treatment. The first 3 patients to complete treatment through week 6 are treated in group A, the next 3 patients in group B, and so on. The treatment period is 4 weeks. Each patient continues on his or her AZT dose as initially administered. The highest dose of AZT that produces less than a 50 percent drop in HIV-1 p24 antigen levels in at least 3 of 5 patients over 6 weeks will be the MED of AZT and will be known as the AZT MED. After the MED is determined, Part 1B begins. Part 1B: 20 patients are randomized to 2 different dosing groups: Group 5: AZT MED (weeks 1 to 8), then AZT MED plus rCD4 (weeks 9 to 16); Group 6: AZT MED plus rCD4 (weeks 1 to 8), then AZT MED (weeks 9 to 16). Part 2: Part 2 begins once accrual to Part 1B is completed. If fewer than 10 of 20 patients exhibit a drop of at least 50 percent in p24 antigen level after receiving AZT and rsCD4 combination treatment, entry to Part 2 will be interrupted and the study design will be reevaluated. In Part 2, 10 patients are randomly assigned to one of four groups. Patients within each group receive two 8 week treatment courses. These two treatment courses are 8 weeks with the AZT MED alone, and 8 weeks of treatment with the combination of the AZT MED plus rCD4.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Nystatin or clotrimazole for suppression of oral thrush.
* Aerosolized pentamidine as chemoprophylaxis for Pneumocystis carinii pneumonia (PCP).
* Trimethoprim / sulfamethoxazole (TMP / SMX) for patients who are clinically and hematologically stable on TMP / SMX PCP prophylaxis.

Patients must have the following:

* Diagnosis of AIDS or advanced AIDS related complex (ARC).
* CD4 cell count < 300 cells/mm3.
* Ability to understand and sign the consent form.

Risk Behavior:

Allowed:

* History of drug abuse with current abstinence or enrollment in a methadone treatment program.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Malignancies other than Kaposi's sarcoma.
* AIDS dementia which, in the opinion of the investigator, precludes patients from giving fully informed consent or from complying fully with the requirements of this protocol.
* Active infection with an opportunistic pathogen requiring ongoing therapy.
* Preexisting antibodies to rCD4.

Concurrent Medication:

Excluded:

* Investigational drugs.
* Antiretroviral agents such as dextran sulfate or AL721.
* Cytotoxic chemotherapy.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Patients with the following are excluded:

* Malignancies other than Kaposi's sarcoma.
* AIDS dementia which, in the opinion of the investigator, precludes patients from giving fully informed consent or from complying fully with the requirements of this protocol.
* Active infection with an opportunistic pathogen requiring ongoing therapy.
* Preexisting antibodies to rCD4.

Prior Medication:

Excluded:

* Zidovudine (AZT) for longer than 30 days or prior treatment with AZT for < 30 days if discontinued for toxicity due to AZT.
* Excluded within 30 days of study entry:
* Immunomodulators.
* Previous participation in any group of another part of this study. For example, patients treated in Part 1A of this study may not reenter the study to be treated in Part 2.
* Chemotherapy.

Prior Treatment:

Excluded within 30 days of study entry:

* Radiation therapy.

Active use of illicit drugs or abuse of alcohol at time of protocol entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Primary Completion 1990-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: RT Schooley, Study Chair; DD Ho, Study Chair; TC Merigan, Study Chair; L Laubenstein, Study Chair
Locations (2):
- United States (2):
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York